CLINICAL TRIAL: NCT06030232
Title: Transarterial Radioembolization (TARE) in COlorectal MEtastasis of Liver
Acronym: TACOME
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Cigdem Soydal, Asc. Prof. of Nuclear Medicine, MD, FEBNM, Ankara University
Other Study IDs: TACOME-TR
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Transarterial Radioembolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observation group: Patients who received radioembolization for colorectal cancer liver metastases
  Interventions: Device: Therasphere

INTERVENTIONS:
Device: Therasphere — Transarterial radioembolization

SUMMARY:
Radioembolization is an established treatment option for patients with unresectable primary and secondary liver tumors. Microspheres containing 90Y are injected intraarterially to deliver a high radiation dose to the tumors. Despite of our knowledge on the effectiveness of 90Y glass microspheres in the treatment of HCC, literature data on the treatment of metastatic colorectal cancer (mCRC) patients with 90Y glass microspheres is limited. In the recent EANM guideline variable healthy liver doses are recommended for patients with mCRC with an effective tumor dose recommendation based on a study with limited number of patients.

Primary objectives; Investigate effective tumor dose and safe healthy liver dose in radioembolization for colorectal cancer liver metastasis using multicompartment dosimetry Secondary objectives; Investigate dose-response and dose-toxicity relationships, time to progress, concordance between pretreatment and posttreatment dose calculations.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* histopathologically proven colorectal cancer diagnosis
* treated with radioembolization for liver metastases with Y90 glass microspheres in lobar or segmental fashion
* have follow-up data at least 6 months after radioembolization

Exclusion Criteria:

* no PET-CT, CT or MR of the liver within last 6 weeks prior to radioembolization.

No PET-CT, CT or MR of the liver 2-4 months after radioembolization Poor image quality Previous local treatment or surgery for the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with metastatic colorectal cancer (mCRC) treated using Y90 glass microspheres in lobar or segmental fashion
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
effective tumor dose and safe healthy liver dose | 3th month after treatment
  Compare the mean effective tumor doses effective tumour dose (in Gy) of patients with or without response to radioembolization for colorectal cancer liver metastasis.

SECONDARY OUTCOMES:
dose (in Gy) -response and dose (in Gy)-toxicity relationships | 6th month after treatment
  Investigate dose-response and dose-toxicity relationships after transarterial radioembolization.

CONTACTS AND LOCATIONS:
Locations (8):
- Turkey (Türkiye) (8):
  - Cukurova University Medical School, Adana
  - Ankara University Medical School, Ankara
  - Hacettepe Univeristy Medical School, Ankara
  - Istanbul University Capa Medical School, Istanbul
  - Istanbul University Cerrahpasa Medical School, Istanbul
  - Marmara University Medical School, Istanbul
  - Yeditepe University Medical School, Istanbul
  - Dokuz Eylul University Medical School, Izmir